CLINICAL TRIAL: NCT01528618
Title: A Randomized, Multicenter Phase III Clinical Trial Comparing Gemcitabine and Cisplatin With 5-Fluorouracil and Cisplatin in the Treatment of Recurrent or Metastatic Nasopharyngeal Carcinoma (NPC)
Brief Title: Effect and Safety Study of GP/FP Regimens in Advanced Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM20110714
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: Advanced Nasopharyngeal Carcinoma; treatment
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Gemcitabine; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gemcitabine and cisplatin (Experimental): gemcitabine 1,000 mg/m2 over 30 to 60 minutes on days 1, 8, and plus cisplatin 80 mg/m2 on day 1, every 3 weeks.
  Interventions: Drug: gemcitabine and cisplatin
- 5-Fluorouracil and cisplatin (Active Comparator): 5-Fluorouracil 4,000 mg/m2 CIV over 96 hours and plus cisplatin 80 mg/m2 on day 1, every 3 weeks.
  Interventions: Drug: 5-Fluorouracil and cisplatin

INTERVENTIONS:
Drug: gemcitabine and cisplatin — The GP regimen consists of gemcitabine at a dose of 1,000 mg/m2 by intravenous (i.v.) infusion over 30 min on day 1 and day 8, and cisplatin 80 mg/m2 by i.v. infusion for 4 h on day 1 only
  Other Names: GP
  Arms: gemcitabine and cisplatin
Drug: 5-Fluorouracil and cisplatin — The FP regimen consists of 5-Fluorouracil 1,000 mg/m2/day which was administered as a continuous intravenous infusion for 96 hours after completion of the cisplatin on days 1( 80 mg/m2 i.v. infusion for 4 h)
  Other Names: FP
  Arms: 5-Fluorouracil and cisplatin

SUMMARY:
The present study will be a randomized, control, multicenter phase III study of recurrent or metastatic (R/M) nasopharyngeal carcinoma (NPC) treated with Gemcitabine (Gemzar, Lilly) and cisplatin regimen (GP) or 5-Fluorouracil plus cisplatin regimen (FP). The population consists of recurrent or metastatic nasopharyngeal carcinoma (NPC) that failed the radical radiotherapy or chemotherapy-naïve advanced NPC (stage IV). The effectiveness and side effects will be evaluated according to Standard WHO response criteria and NCI-CTC AE V3.0.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is most commonly seen in Southeast Asia, especially in southern and southeastern China ,where the incidence rate has been documented between 10 and 150 cases per 100,000 population per year. NPC is a radiosensitive tumor, and radiotherapy is considered to be the treatment of choice for most cases. The 5-year survival rate (all stages) is around 50% .In other words, more than half of the NPC cases will eventually fail radiotherapy and reasons of the failure are both local relapse and remote metastasis.

For these advanced or metastatic NPC, chemotherapy is the most important therapeutics,and they are relatively responsive to chemotherapy compared to other head and neck cancers. The backbone of the treatment for recurrent/metastatic (R/M) NPC is cisplatin containing regimen, which is also regarded as the standard regimen for other squamous cell carcinoma of head and neck (SCCHN). The FP regimen is widely used in R/M NPC patients now and its response rate is around 40%-65%,but the response period is usually short and the adverse reaction is frequent and badly tolerant, which influent the treatment compliance seriously. What's more, the catheters and pumps are necessary for continuous infusion of 5-Fluorouracil, which add to the cost, immobility and inconvenience of the treatment.

Preclinical and clinical data show synergistic activity between gemcitabine and cisplatin without overlapping toxicity. Several clinical trials enrolling a minority of advanced NPC patients suggest GP regimen has promising effectiveness and well tolerated side effects, and they indicated a potential possibility that the GP regimen comes to the standard first line choice instead of the FP regimen

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NPC diagnosis
* Elder than 18 years old are inclusive
* Recurrence or metastatic nasopharyngeal carcinoma with evidence of unsuitable for local treatment
* Amenable to regular follow-up
* Subjects with at least one measurable lesion (Tumor lesions that are situated in a previously irradiated area could not be considered measurable).
* Performance status: 0-1(ECOG)
* WBC > 4.0X109/L, PLT > 100X109/L, with normal hepatic function(AST, ALT < 2.5 x upper limit of normal , and bilirubin < 1.5 x upper limit of normal), with normal renal function (Creatinine < 1.5 x upper limit of normal)
* No chemotherapy or radical radiotherapy received within 6 months prior to enrollment
* Life expectancy over twelve weeks
* Signed and dated informed consent before the start of specific protocol procedures
* Ability to comply with trial requirements.

Exclusion Criteria:

* Patient suitable for local treatment (eg. radiotherapy)
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* Patient with central nervous system metastasis
* Patient life threatening medical condition
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and two weeks after the completion of trial.
* Performance status ≥ 2
* With a pre-existing peripheral neuropathy (National Cancer Institute Common Toxicity Criteria for Adverse Events [NCI CTC] grade ≥ 2)
* Serious concurrent illness
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors[Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
* Patient refusing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2012-02-21 (Actual); Primary Completion 2016-04-10 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) assessed by independent image committee and the investigators | 36 months

SECONDARY OUTCOMES:
Overall survival (OS) | 36 months
Objective response rate (ORR) | 36 months
Number of Participants with Adverse Events | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: li zhang, doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Medical Oncology,Cancer Center of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Hong S, Zhang Y, Yu G, Peng P, Peng J, Jia J, Wu X, Huang Y, Yang Y, Lin Q, Xi X, Xu M, Chen D, Lu X, Wang R, Cao X, Chen X, Lin Z, Xiong J, Lin Q, Xie C, Li Z, Pan J, Li J, Wu S, Lian Y, Yang Q, Zhao C, Fang W, Zhang L. Gemcitabine Plus Cisplatin Versus Fluorouracil Plus Cisplatin as First-Line Therapy for Recurrent or Metastatic Nasopharyngeal Carcinoma: Final Overall Survival Analysis of GEM20110714 Phase III Study. J Clin Oncol. 2021 Oct 10;39(29):3273-3282. doi: 10.1200/JCO.21.00396. Epub 2021 Aug 11. PMID 34379443
- [Derived] Zhang L, Huang Y, Hong S, Yang Y, Yu G, Jia J, Peng P, Wu X, Lin Q, Xi X, Peng J, Xu M, Chen D, Lu X, Wang R, Cao X, Chen X, Lin Z, Xiong J, Lin Q, Xie C, Li Z, Pan J, Li J, Wu S, Lian Y, Yang Q, Zhao C. Gemcitabine plus cisplatin versus fluorouracil plus cisplatin in recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2016 Oct 15;388(10054):1883-1892. doi: 10.1016/S0140-6736(16)31388-5. Epub 2016 Aug 23. PMID 27567279